CLINICAL TRIAL: NCT05535673
Title: A Single Dose-escalation Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Allogeneic CAR-T Targeting CD19 in Patients With Refractory or Relapsed B Cell Lymphoma
Brief Title: Safety, Efficacy and Pharmacokinetics of ThisCART19A in Patients With Refractory or Relapsed B Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhengzhou University (Other)
Collaborators: Fundamenta Therapeutics, Ltd. (Industry)
Responsible Party: Principal Investigator, Mingzhi Zhang, Principal Investigator, Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT400-010
Record Dates: First submitted 2022-08-30; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Allogeneic, CAR-T, Protein Sequestration, Non-gene Edited, r/r B-NHL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART19A cell injection (Experimental): In this study, allogeneic anti-CD19 CART cell (This CART19A) injection is used to treat patients with refractory or relapsed CD19 positive B cell Lymphoma.
  Interventions: Drug: ThisCART19A

INTERVENTIONS:
Drug: ThisCART19A — In this study, allogeneic anti-CD19 CAR-T cell (ThisCART19A) injection is used to treat patients with refractory or relapsed CD19 positive B cell Lymphoma.

SUMMARY:
This is a single dose escalation study to evaluate the safety, efficacy and pharmacokinetics of ThisCART19A (Allogeneic CAR-T targeting CD19) in patients with refractory or relapsed CD19 positive B cell Lymphoma.

DETAILED DESCRIPTION:
This is a single-center, nonrandomized, open-label, dose-escalation study to evaluate the safety, efficacy and pharmacokinetics of ThisCART19A in patients with refractory or relapsed CD19 positive B cell Lymphoma, such as Diffuse large B-cell lymphoma (DLBCL) , follicular lymphoma and etc.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years old;
2. Histologically confirmed diagnosis per WHO Classification Criteria for Lymphocytic Tumors 2017, including follicular lymphoma (FL), marginal zone lymphoma (MZL, including SMZL, NMZL and extranodal MZL), mantle cell lymphoma (MCL), diffuse large B-cell lymphoma (DLBCL), etc;
3. Relapsed or refractory B-cell NHL.
4. Adequate treatment :

   1. Follicular lymphoma should be treated with at least two prior treatment including alkylating agents and anti-CD20 mAbs;
   2. Marginal zone lymphoma should be treated with at least two prior treatment including anti-CD20 mAbs;
   3. mantle cell lymphoma should be treated with a first-line therapy including anthracyclines/bendamoxetine+anti-CD20 mAbs;
   4. Diffuse large B lymphoma, not otherwise specified (DLBCL, NOS), high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (double/triple hit lymphoma, DHL/THL), diffuse large B-cell lymphoma (DLBCL) transformed from follicular lymphoma (FL), histological grade 3b follicular lymphoma. relapsed or primary refractory lymphoma within 12 months after first-line treatment, first-line therapy including anthracycline and anti-CD20 mAbs.
5. Failing to autologous CAR-T therapy.
6. Estimated life expectancy > 12 weeks deemed by investigator；
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
8. At least one measurable lesion, with any nodal lesion > 15mm in the longest diameter and any extranodal lesion > 10mm in the longest diameter.
9. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function;
10. Should be confirmed Cluster of differentiation(CD)19 positive by biopsy for the patient who received target CD19 therapy before.

Exclusion Criteria:

1. Allergic to preconditioning measures.
2. HP-positive MALT;
3. Patients with risks of deep gastrointestinal ulcers, perforation or gastrointestinal bleeding
4. Patients with other malignancies other than B-cell malignancies within 5 years prior to screening. Patients with cured skin squamous carcinoma, basal carcinoma, non-primary invasive bladder cancer, localized low-risk prostate cancer, in situ cervical/breast cancer can be recruited.
5. Uncontrollable bacterial, fungal and viral infection during screening.
6. Patients had pulmonary embolism (PE) and/or deep vein thrombosis (DVT) within 3 months prior to enrollment.
7. Had intolerant severe cardiovascular and cerebrovascular diseases and hereditary diseases prior to enrollment.
8. Imaging confirmed the presence of central nervous system involvement (both primary and secondary) and obvious symptoms at the time of screening.
9. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) or Human immunodeficiency virus (HIV) or Syphilis infection. HBV-DNA < 2000 IU/mL can be enrolled, but should admitted to use anti-virus drugs such as entecavir, tenofovir, etc, and supervisory the relative indication during the treatment.
10. Had big lesion(single lesion diameter ≥7.5 cm).
11. Receive allogeneic hematopoietic stem cell transplantation less than 100 days.
12. Vaccinated with influenza vaccine within 2 weeks prior to lymphodepleting chemotherapy (Severe Acute Respiratory Syndrome-Corona virus disease 19 can be included, inactivated, live/non-live adjuvant vaccinations allowed to be included) .
13. Patients who are receiving Graft versus host disease Hepatitis(GvHD) treatment; Patients without GvHD and who had stopped immunosuppressive drugs for at least 1 month were eligible for inclusion.
14. Women who are in pregnant or lactating, and female subjects or partners who plan to be pregnant within 1 year after cell infusion. Male subjects who plan pregnancy within 1 year after infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-02 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) observation in patient with NHL during dose escalation stage | 28 days
  DLT is defined as the incidence of severe adverse events related to ThisCART19A more than 33% in each dose level.
The incidence of all grade TEAEs and ≥3 grade TEAEs during dose escalation stage | Up to 2 years after ThisCART19A infusion
  Incidence of treatment-emergent adverse events (TEAEs) and ≥3 grade TEAEs
Objective Response Rate in patient with NHL during dose expansion stage | 12 months
  the incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as best response to treatment

SECONDARY OUTCOMES:
Analysis the severity and Incidence of Adverse Events in each dose level during dose escalation and dose expansion stage | 3 months
  Including more than or equal to grade 3 adverse events graded according to the NCI CTCAE v5.0, or the adverse events with special attention
Analysis the change characteristics of CART cell number and copy number during dose escalation and expansion stages | 6 months
  Track CAR T cells expansion in patients after infusion
the change characteristics of immune effect cells number during dose escalation and expansion stages | 3 months
  Analysis the effect cells (such as CD19+ B cells、T cells、NK cells)
Analysis the change characteristics of cytokines during dose escalation and expansion stages (IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12p70/IL-17A/IL-17F/IL-22/TNF-α/TNF-β) | 3 months
  cytokines including IL-1β/IL-2/IL-4/IL-5/IL-6/IL-8/IL-10/IL-12p70/IL-17A/IL-17F/IL-22/TNF-α/TNF-β
Duration of response (DOR) during dose escalation stage and expansion stage | 12 months
  The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR)
Progress-free survival (PFS) during dose escalation stage and expansion stage | 12 months
  Progress-free survival (PFS) is defined as time from the first CAR-T cell infusion date to first documentation of PD, or death from any cause.
OS(overall survival) during dose escalation stage and expansion stage | 12 months
  Overall survival (OS) is defined as the time from the date of lymphodepletion until death from any cause.

IPD SHARING:
Plan to Share IPD: No